CLINICAL TRIAL: NCT03757520
Title: Evaluation of Text Neck Syndrome and Hand Grip Force in Smart Phone Addiction Among Students of Jazan University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wafaa Mahmoud Amin (Other Government)
Responsible Party: Sponsor-Investigator, Wafaa Mahmoud Amin, Principal Investigator, University of Jazan
Organization: University of Jazan (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 0018827704
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Pain, Back; Neck Pain; Postural; Strain; Myofascial Pain Syndrome
MeSH Terms: conditions — Back Pain; Neck Pain; Sprains and Strains; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: According two Smartphone Addiction Proneness Scale (SAPS) the subjects will be divided into two groups: Regular user group with SAPS score 39 or less. Heavy user group with SAPS score 40 or more.
  we have two variables to be assessed:
  1. Pain pressure threshold for two muscles (upper fiber of trapezius and sternocleidomastoid muscle)
  2. Hand grip force
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular user group (Active Comparator): Their number: 300; female and male students, will earn 39 points or less of Smartphone Addiction Proneness Scale. Pain Pressure Threshold and Hand Grip Force will Measured for them.
  Interventions: Diagnostic Test: Pain Pressure Threshold; Diagnostic Test: Hand Grip Force
- Heavy user group (Active Comparator): Their number: 300; female and male students, will earn 40 points or more of Smartphone Addiction Proneness Scale. Pain Pressure Threshold and Hand Grip Force will Measured for them.
  Interventions: Diagnostic Test: Pain Pressure Threshold; Diagnostic Test: Hand Grip Force

INTERVENTIONS:
Diagnostic Test: Pain Pressure Threshold — The pain pressure thresholds (PPTs) will be measured using an pressure algometer commander over potential trigger points (TrPs) on the body for upper fiber of trapezius, and sternocleidomastoid muscle.
  Other Names: PPTs
Diagnostic Test: Hand Grip Force — For measuring the grip strength, the subjects will be asked to sit on a chair with their hip joint flexed at 90 degree, and shoulder joint in a neutral position.
  The elbow is fixed at 90 degree flexion, forearm in a neutral position, and wrist at 0 to 15 degree radial deviation The test will be performed twice, and the higher value between the two measurements will be selected.

SUMMARY:
This study will be conducted in the Department of physical therapy, College of Applied Medical Sciences,Jazan University, to investigate text neck syndrome and hand grip force in smart phone addiction among students of jazan university

DETAILED DESCRIPTION:
Four hundreds students with age 19 to 26 years old, and right dominant hand, will be recruited from the College of Applied Medical Sciences, Jazan University. Subjects will be randomly assigned to into a heavy user group (n=300; female and male students) and a control or regular use group (n=300; female and male students) according to their smartphone addiction proneness scale.

Baseline hydraulic hand dynamometer: (Fabrication Enterprises Incorporated, White Plains,New York, USA) is used to measure the hand grip strength and pinch strength.

Algometer Commander (JTech Medical Company) is used on the location of the trigger point to assess the amount of pressure the patient could sustain before the patient registered the pressure as being painful for upper fiber of trapezius muscle and sternocleidomastoid muscle

ELIGIBILITY:
Inclusion Criteria:

1. The participant will be right-handed.
2. No abnormal findings confirmed through physical and neurological examination.
3. No congenital abnormalities in either the cervical or the lumbar spine.
4. No history of severe surgical procedures ( Park et al., 2015) .

Exclusion Criteria:

1. History of a neurological disease.
2. History of musculoskeletal injury of neck and lumbar region.
3. Unstable medical condition.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2019-08-11 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold for upper fiber of trapezius muscle | 3 minutes
  Using Algometer to measure pain pressure for upper trapezius trigger point which lies in the more horizontal fibers of the upper trapezius on the back of the shoulder, about halfway between spine and the acromion on right and left side for 3 repetition for each
Pain pressure threshold for sternocleidomastoid muscle | 9 minutes
  Using Algometer to measure pain pressure for sternocleidomastoid muscle on right and left side for 3 repetition for each. Measurement will includes three sites on each side:
  1. upper part of the sternal division of the muscle near to its insertion into the mastoid process. 2. he mid-part of the sternal division of the muscle. 3. lower end of this division near to its attachment to the sternum.
Hand Grip Force | 15 minutes
  For measuring the grip strength, the subjects will be asked to sit on a chair with their hip joint flexed at 90 degree, and shoulder joint in a neutral position.
  The elbow is fixed at 90 degree flexion, forearm in a neutral position, and wrist at 0 to 15 degree radial deviation.The test will be performed twice, and the higher value between the two measurements will be selected.
  The subjects are allowed a rest time of more than 5 minutes after the first measurement to avoid examiner bias and to decrease physical stress

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
there is no plan